CLINICAL TRIAL: NCT01410305
Title: Vitamin D Metabolism Inflammation, and Cardiovascular Risk in HIV-infected Children and Young Adults
Brief Title: Vitamin D and HIV-Cardiovascular Disease in Children and Young Adults
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Emory-Children's Center (Other)
Responsible Party: Principal Investigator, Grace McComsey, Professor of Pediatrics and Medicine, University Hospitals Cleveland Medical Center
Other Study IDs: 1R01HD070490-01 (NIH)
Record Dates: First submitted 2011-08-04; First posted 2011-08-05 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D Deficiency; HIV+ Children; HIV+ Young Adults
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, serum, PBMCs, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV+: HIV Positive children or young people between the ages of 8 and 25
- HIV Negative: HIV Negative matched controls by age and race

SUMMARY:
The relationship of Vitamin D levels in children and young adults to atherosclerosis.

ELIGIBILITY:
Inclusion Criteria - Documentation of HIV Infection Between ages of 8 and 25

* On stable ART for at least 12 weeks for the HIV+ patients
* Cumulative duration of ART for at least 48 weeks for HIV + patients
* Healthy child/young adult with age and race matched to HIV+ patient for the HIV- controls
* Absence of HIV based on medical and medication history

Exclusion Criteria:

* Taking > 800 IU of Vitamin D per day
* Parathyroid or Calcium disorders
* Acute illness and active inflammatory condition
* Chronic illnesses that include malignancy, diabetes, CAD
* Pregnancy and lactation
* Creatinine Clearance <50 ml/min
* Hgb < 9.0 g/dL
* AST and ALT > 2.5 upper limits of normal

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Any HIV+ patient between the ages of 8 and 25 and matched HIV- controls matched by age and race.
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2011-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Vitamin D levels | One time point at entry
  To perform a cross-sectional analysis of blood vitamin D status among the HIV-infected children and young adults to evaluated the point prevalence fo plasma 25(OH)D levels indicating vitamin D insufficiency, deficiency and severe deficiency, and to compare the prevalence to a matched uninfected healthy control group.

CONTACTS AND LOCATIONS:
Overall Officials: Grace McComsey, MD, Principal Investigator — University Hospitals Cleveland Medical Center; Allison Ross Eckard, MD, Principal Investigator — Emory-Children's Center
Locations (2):
- United States (2):
  - Emory Chldren's Center, Atlanta, Georgia
  - University Hospitals Case Medical Center, Case Western Reserve University, Cleveland, Ohio